CLINICAL TRIAL: NCT01221675
Title: Prospective Multicentric Optimization and Phase I/II Study of Pretargeted Radioimmunotherapy (PRAIT) Using Anti-CEA x Anti-HSG TF2 Bispecific Antibody (bsMAb) and 177Lu-IMP-288 Peptide in Patients With CEA-expressing Small Cell Lung Carcinoma (SCLC) or CEA-expressing Non Small Cell Lung Carcinoma (NSCLC)
Brief Title: TF2- Small Cell Lung Cancer Radio Immunotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre René Gauducheau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 08/9-O
Record Dates: First submitted 2010-10-11; First posted 2010-10-15 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-04

CONDITIONS: Small Cell Lung Cancer; CEA-expressing Non Small Cell Lung Carcinoma (NSCLC)
Keywords: Small Cell Lung Cancer or CEA-expressing Non Small Cell Lung Carcinoma (NSCLC); Radio Immunotherapy; Lutetium; patient ≥ 18 years of age with CEA-positive SCLC in partial response; or who failed at least two lines of standard radiation and/or chemotherapy; or Patients with histologic diagnosis of NSCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Antibody TF2 — preciblage with an antibody
Radiation: IMP-288-Lutetium — Internal Radiation
Radiation: IMP-288-Indium — Imaging

SUMMARY:
Lung cancer is currently the leading cause of cancer death in both men and women in Europe, with an estimated 250000 new cases diagnosed in 2005. The continued poor outcome of patients indicates that the current recommended regimens are falling short. In addition, many of the commonly used chemotherapy agents are associated with severe nonhematologic toxicities that are often cumulative and nonreversible and impair quality of life in this essentially palliative setting. Therefore, agents with novel mechanisms of action and superior safety profiles need to be investigated. More than 50% of lung cancer shows carcinoembryonic antigen (CEA) expression and anti-CEA radioimmunotherapy (RAIT) could be used. The investigators group showed that pretargeted RAIT (PRAIT) using bispecific antibody (bsMAb) can deliver a higher radiation dose to a tumor than a directly radiolabeled anti-CEA antibody, and shows improved anti-tumor efficacy. This clinical trial is designed to assess PRAIT using an entirely new recombinant anti-CEA bsMAb and a 177Lu-labeled peptide for the treatment of CEA-expressing small cell lung cancers (SCLC) or CEA-expressing Non Small Cell Lung Carcinoma (NSCLC)

DETAILED DESCRIPTION:
The purpose of this open-label prospective optimization and phase I/II clinical trial is to examine the safety, optimal dose, targeting, dosimetry and efficacy of PRAIT using the humanized anti-CEA x anti-HSG bsMAb TF2 and the 177Lu-IMP-288 peptide pretargeted in patients with CEA-positive SCLC or CEA-expressing Non Small Cell Lung Carcinoma (NSCLC)

This study has 2 parts: Study plan I (Optimization study) and Study plan II (Escalating activity phase I/II study).

The Study plan I is designed to optimize the pretargeting procedure using blood pharmacokinetics (Pk) and dosimetry in 9 patients receiving escalating doses of TF2 followed 2 to 4 days later by 1.1 GBq/m2 of 177Lu-IMP-288.

The study plan II is designed to determined MTD of 177Lu-IMP-288 using dosimetry and toxicity data in a phase I/II study performed in patients receiving optimal dose of TF2 bsMAb (determined in study plan I) followed 2 to 4 days by escalating activity of 177Lu-IMP-288.

A pre-therapy imaging study (using TF2 followed 2 to 4 days later by 185 MBq of 111In-IMP-288) is performed in the two study plans to qualify a patient for treatment with the subsequent therapy dose.

ELIGIBILITY:
Inclusion Criteria:

• Patients with histologic diagnosis of SCLC who are in partial response or who have failed at least two lines of standard radiation and/or chemotherapy. Outside formal contra-indication, patients must have received at least one prior platinum-based chemotherapy.

or

* Patients with histologic diagnosis of NSCLC (without activating mutation of EGFR gene) who have failed at least one line of chemotherapy (platinum in combination with a third generation drug or combination of 2 third generation drug +/-bevacizumab in case of predominance of non-squamous tumor)
* Age ≥ 18 years
* At least 4-weeks after the previous treatment and have recovered from previous radio- or chemotherapy
* Women of child-bearing potential must have a negative pregnancy test.
* Karnofsky performance status ≥ 60 or ECOG performance status 0-2Karnofsky
* Minimum life expectancy of 3 months
* Positive CEA on immunohistology or plasma CEA ≥ 10 ng/mL
* At least one measurable lesion by CT
* At least one abnormal focus by FDG-PET
* Imaging studies must be performed within 1-4 weeks before PRAIT study to document extent of disease
* Signed informed consent form.

Exclusion Criteria:

* Pregnant or lactating woman. Women of child-bearing potential will be asked to practice adequate means of birth control for a minimum of 12 months after treatment.
* Male patient refusing effective contraception for a minimum of 12 months after treatment.
* Brain metastases but patients with brain metastases controlled after treatment by Surgery or radiotherapy since more than 4 weeks are eligibles for the study. An treatment by associated corticotherapy is authorized for these patients.
* Known HIV or hepatitis
* Any serious active disease or comorbid medical condition (according to the investigator's decision and information provided in the IDB)
* Severe disorders of hemostasis or anticoagulant treatment cure
* Extensive irradiation to more than 25% of their red marrow
* Bone marrow involvement to more than 25%
* External radiation to specific organs or areas at the maximum tolerated level
* EGFR gene mutation in tumor (only for NSCLC)
* Febrile aplasia during a previous chemotherapy
* Neutrophils < 1.5 G/l
* Platelets < 100 G/l
* Uncontrolled diabetes
* Poor renal function (creatinine level > 2.5 maximum normal level)
* Poor hepatic function (total bilirubin level > 30 mmol/l, transaminases > 2.5 maximum normal level)
* Treatment with any investigational drug within 30 days before planned PRAIT and during the study
* Any history of cancer during the last 5 years, with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma,
* Presence of anti-antibody reactivity
* Known hypersensitivity to murine antibodies or proteins
* Adult patient unable to give informed consent because of intellectual impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint of study plan I: To determine the optimal TF2 protein dose for pretargeting IMP-288.
Primary endpoint of study plan II • the maximum tolerated dose (MTD) for the TF2-pretargeted 177Lu-IMP-288 under optimal pretargeting conditions.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU d'Angers, Angers
  - CHU, Brest
  - Centre Jean Perrin, Clermont-Ferrand
  - Hôpital La tronche, Grenoble
  - Hotel Dieu, Nantes
  - Centre René Gauducheau, Saint-Herblain

REFERENCES:
- [Derived] Bodet-Milin C, Ferrer L, Rauscher A, Masson D, Rbah-Vidal L, Faivre-Chauvet A, Cerato E, Rousseau C, Hureaux J, Couturier O, Salaun PY, Goldenberg DM, Sharkey RM, Kraeber-Bodere F, Barbet J. Pharmacokinetics and Dosimetry Studies for Optimization of Pretargeted Radioimmunotherapy in CEA-Expressing Advanced Lung Cancer Patients. Front Med (Lausanne). 2015 Nov 27;2:84. doi: 10.3389/fmed.2015.00084. eCollection 2015. PMID 26640780